CLINICAL TRIAL: NCT04487899
Title: Analysis of Heart Rate Variability During Emergency Flight Simulator Missions in Fighter Pilots
Status: Completed | Type: Observational
Sponsor: Universidad de Extremadura (Other)
Responsible Party: Principal Investigator, Carlos Fernández-Morales, Principal Investigator, Universidad de Extremadura
Other Study IDs: 02
Record Dates: First submitted 2020-07-22; First posted 2020-07-27 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-09

CONDITIONS: Heart Rate Variability; Autonomic Nervous System
Keywords: Emergency missions; Assesment; Military Health Services; heart rate variability; autonomic nervous system

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Instructors group: Group of flight instructors at the reactor school.
  Interventions: Device: Analysis of heart rate variability
- Students group: Group of students at the reactor school.
  Interventions: Device: Analysis of heart rate variability

INTERVENTIONS:
Device: Analysis of heart rate variability — The HR HRV interval of the heartbeat (variations in the time interval between beats) was used as a measure of autonomous modulation, and the Firstbeat Bodyguard monitor (Firstbeat Technologies, Jyväskylä, Finland) was used to record HRV data during the session with emergency situations in the flight simulator. Data was downloaded from the devices to a computer using Firstbeat Uploader software (Firstbeat Technologies), and all R-R interval series were imported into the Kubios software package (University of Eastern Finland, Kuopio, Finland). To calculate the autonomous equilibrium, the commonly used HRV method based on the Poincaré graph was used (Brennan et al., 2001; Mourot et al., 2004).

SUMMARY:
The autonomous response of fighter and attack pilots who attend sessions in a flight simulator will be evaluated by measuring and analyzing heart rate variability (HRV).

DETAILED DESCRIPTION:
The autonomous response of fighter and attack pilots during emergency situations in a flight simulator will be assessed by measuring and analysing heart rate variability (HRV). Eighteen pilots with instructor or student status assigned at the time of the evaluation to the ALA 23 district of the Talavera la Real Air Base of the Ministry of Defence of the Spanish Government (Badajoz) were studied during emergency situations in flight simulator. Subjects were assigned by non-probabilistic randomisation to an instructor group (IG; 7 subjects), and to a student group (AG; 11 subjects).

The recording of the parameters indicated corresponds to the emergency situations described above. Data collection was made in three different moments:

1. Take-off: it starts after reading the checklist until the engine fault is resolved.
2. Flight: during manoeuvres characterised by the recovery of abnormal positions.
3. Landing: where the pilot performs the landing manoeuvre, with the loss of spatial situation.

ELIGIBILITY:
Inclusion Criteria:

* Pilots who had the status of instructor or student assigned at the time of assessment to the ALA 23 district of the Talavera la Real Air Base of the Ministry of Defense of the Government of Spain (Badajoz).

Exclusion Criteria:

* Any uncontrolled neurological or cardiac disorder.
* Being involved in ongoing medical-legal conflicts.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The selection of the sample was made in the accessible population of the Talavera la Real Air Base (Badajoz).
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2019-11-18 (Actual); Study Completion 2020-03-10 (Actual)

PRIMARY OUTCOMES:
Root Mean Square of the Successive Differences (RMSSD) | 1 week
  It indicates the degree of activation of the Parasympathetic Nervous System on the cardiovascular system. It is obtained from the square root of the mean value of the sum of the squared differences of all successive RR intervals. This parameter reports the short-term variations of the RR intervals. It is directly associated with short-term variability.
Stress Score | 1 week
  It is an index described by Naranjo-Orellana et al. to facilitate physiological interpretation of Poincaré plot. It is expressed as the inverse of the SD2 diameter multiplied by 1000 and is considered directly proportional to the sympathetic activity in the sinus node.
Sympathetic/parasympathetic ratio (S/PS) | 1 week
  It is also described by Naranjo-Orellana et al., S/PS is expressed as the quotient of SS and SD1, and it is considered to reflect autonomic balance - that is, the relationship between sympathetic and parasympathetic activity

SECONDARY OUTCOMES:
Standard Deviation 1 (SD1) | 1 week
  It indicates the sensitivity of short-term variability in HRV non-linear spectrum. It is considered an indicator of parasympathetic activity.
Standard Deviation 2 (SD2) | 1 week
  It is a diameter from Poincaré plot which indicates the degree of longitudinal dispersion. It is thought to reflect long-term changes in RR intervals and it is considered an inverse indicator of parasympathetic activity.
Min_HR | 1 week
  Minimum heart rate variability.
Max_HR | 1 week
  Maximum heart rate variability.
Mean_HR | 1 week
  It corresponds to the interval between two beats (R peaks on the ECG).
pNN50 | 1 week
  Percentage of consecutive RR intervals that differ by more than 50 ms from each other. A high value of pNN50 provides valuable information about high spontaneous HR.
Low Frequency Power (LF) | 1 week
  Situated between 0.04 and 0.15 Hz. In long-term recordings it provides us with more information about the activity of the SNS.
High Frequency Power (HF) | 1 week
  They are located between 0.15 and 0.4 Hz. HF is clearly related to PNS activity and has a relaxation-related effect on HR2.
Low/High Frequency ratio (HF/LF) | 1 week
  From low frequency and high frequency ratio of the HRV spectral analysis result we can estimate the vagal (related to relaxation and HF) and sympathetic (related to stress and LF) influence. Thus we can estimate sympathetic-vagal balance.

CONTACTS AND LOCATIONS:
Overall Officials: Luis Espejo-Antúnez, PhD, Principal Investigator — Universidad de Extremadura
Locations (1):
- Universidad de Extremadura, Badajoz, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] de la Cruz Torres B, Albornoz Cabello M, Garcia Bermejo P, Naranjo Orellana J. Autonomic responses to ultrasound-guided percutaneous needle electrolysis of the patellar tendon in healthy male footballers. Acupunct Med. 2016 Aug;34(4):275-9. doi: 10.1136/acupmed-2015-010993. Epub 2016 Jan 20. PMID 26792776
- [Background] Kitagawa Y, Kimura K, Yoshida S. Spectral analysis of heart rate variability during trigger point acupuncture. Acupunct Med. 2014 Jun;32(3):273-8. doi: 10.1136/acupmed-2013-010440. Epub 2014 Mar 7. PMID 24610637
- [Background] Mourot L, Bouhaddi M, Perrey S, Rouillon JD, Regnard J. Quantitative Poincare plot analysis of heart rate variability: effect of endurance training. Eur J Appl Physiol. 2004 Jan;91(1):79-87. doi: 10.1007/s00421-003-0917-0. Epub 2003 Sep 4. PMID 12955518
- [Background] Gil-Rodas F, Pedret C, Ramos-Castro J, Capdevila-Ortís L. Variabilidad de la frecuencia cardíaca: concepto, medidas y relación con aspectos clínicos (I). Arch Med Deporte Rev Fed Esp Med Deporte Confed Iberoam Med Deporte. 2008;(123):41-8.
- [Background] Malik M. Heart rate variability: Standards of measurement, physiological interpretation, and clinical use: Task force of the European Society of Cardiology and the North American Society for Pacing and Electrophysiology. Ann Noninvasive Electrocardiol. 1996;1(2):151-81.
- [Background] Naranjo Orellana J, de la Cruz Torres B, Sarabia Cachadina E, de Hoyo M, Dominguez Cobo S. Two new indexes for the assessment of autonomic balance in elite soccer players. Int J Sports Physiol Perform. 2015 May;10(4):452-7. doi: 10.1123/ijspp.2014-0235. Epub 2014 Oct 29. PMID 25364865
- [Derived] Fernandez-Morales C, Espejo-Antunez L, Clemente-Suarez VJ, Tabla-Hinojosa FB, Albornoz-Cabello M. Analysis of heart rate variability during emergency flight simulator missions in fighter pilots. BMJ Mil Health. 2024 Jul 24;170(4):296-302. doi: 10.1136/military-2022-002242. PMID 36585028